CLINICAL TRIAL: NCT04813952
Title: The Effect of Minimal Flow Sevoflurane Anesthesia on Blood Gas Analysis and Hemodynamic Parameters in Laparoscopic Cholecystectomies, a Randomised Controlled Trial.
Brief Title: The Effect of Minimal Flow Sevoflurane Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nebia Peker, medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1019
Record Dates: First submitted 2021-03-10; First posted 2021-03-24 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Anesthesia; Functional; Anesthesia Awareness
Keywords: minimal flow anesthesia; laparoscopic cholecystectomy
MeSH Terms: conditions — Intraoperative Awareness | interventions — Sevoflurane

STUDY DESIGN:
Intervention Model Description: they will divided into two equal groups as Group M (minimal flow anesthesia group) with fresh gas flow 0,5 L.min-1 and Group C (high flow anesthesia/ control group) with fresh gas flow 4 L.min-1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group M (Active Comparator): Group M is minimal flow anesthesia group with fresh gas flow 0,5 L.min-1. Thirty five patients with ASA class I-II and between the ages of 18-65 undergoing elective laparoscopic cholecystectomy will be included. These patients were planned to be administered sevoflurane anesthesia with 0,5 L.min-1 flow under general anesthesia.
  Interventions: Drug: Sevoflurane inhalant product
- Group H (Active Comparator): Group H is high flow anesthesia group with fresh gas flow 4 L.min-1. Thirty five patients with ASA class I-II and between the ages of 18-65 undergoing elective laparoscopic cholecystectomy will be included. These patients were planned to be administered sevoflurane anesthesia with 4 L.min-1 flow under general anesthesia.
  Interventions: Drug: Sevoflurane inhalant product

INTERVENTIONS:
Drug: Sevoflurane inhalant product — The sevoflurane dose differed in both groups in relation to the fresh gas flow. Since the fresh gas flow is less in group M, the concentration of sevoflurane consumed by the patient at the end of the case will be less.
  Other Names: Sevorane

SUMMARY:
Our aim is to investigate the effect of minimal flow anesthesia with sevoflurane on hemodynamics and arterial blood gas parameters in laparoscopic cholecystectomy operations.

DETAILED DESCRIPTION:
Introduction: Low-flow anesthesia techniques have regained popularity in recent years with the development of low solubility volatile agents such as sevoflurane and desflurane, and modern anesthesia devices. Reducing the flow of fresh gas as much as possible will reduce the amount of volatile agent used, thus preventing air pollution, providing lower costs, and also preserving heat and moisture in the respiratory tract by using rebreathing systems. Laparoscopic surgery is superior to open surgical techniques due to its minimally invasive nature, less postoperative pain, less incidence of wound infections, shortening the hospitalization, and allowing patients to return to their normal lives sooner after the operation.

Our aim is to investigate the effect of minimal flow anesthesia with sevoflurane on hemodynamics and arterial blood gas parameters in laparoscopic cholecystectomy operations.

Material and Method: Seventy patients with ASA (American Society of Anesthesiologists) class I-II between the ages of 18-65 undergoing elective laparoscopic cholecystectomy were included in the study. After the patients were randomly selected by computer, they were divided into two equal groups as Group M (minimal flow anesthesia group) with fresh gas flow 0,5 L.min-1 and Group C (high flow anesthesia/ control group) with fresh gas flow 4 L.min-1. In both groups. Demographic data, duration of anesthesia, operation times, recovery times, hemodynamic parameters and arterial blood gas parameters of all patients were recorded. The patient data collected in both groups were compared statistically.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) class I-II
* The operation time between 60-180 minutes

Exclusion Criteria:

* Severe cardiac disease
* COPD (Chronic Obstructive Pulmonary Disease)
* Severe liver and kidney disease,
* Diabetes mellitus
* Morbid obesity
* Alcohol and/or drug addiction
* Risk or history of malignant hyperthermia
* Pregnancy and lactation
* Emergency cases
* Operation time less than 60 minutes and longer than 180 minutes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
CHANGE IN P/F | from the beginning to the end of anesthesia
  PaO2/FiO2 ratio is the ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2 expressed as a fraction, not a percentage). P/F ratio is a widely used clinical indicator of hypoxaemia
CHANGE IN PaCO2 | from the beginning to the end of anesthesia
  The partial pressure of carbon dioxide is the measure of carbon dioxide within arterial blood.

SECONDARY OUTCOMES:
volatile agent consumption amount | from the beginning to the end of anesthesia
  the total amount of volatile agent (sevoflurane) consumed at the end of the surgery

OTHER OUTCOMES:
CHANGE IN HR | from the beginning to the end of anesthesia
  Heart rate per minute
CHANGE IN MAP | from the beginning to the end of anesthesia
  Mean arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Nurcan Coşkun, Study Chair — Sisli Hamidiye Etfal Training and Research Hospital; Serkan İslamoğlu, Study Chair — Sisli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Nebia Peker, Şişli, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Doger C, Kahveci K, Ornek D, But A, Aksoy M, Gokcinar D, Katar D. Effects of Low-Flow Sevoflurane Anesthesia on Pulmonary Functions in Patients Undergoing Laparoscopic Abdominal Surgery. Biomed Res Int. 2016;2016:3068467. doi: 10.1155/2016/3068467. Epub 2016 Jun 20. PMID 27413741
- [Result] Park SY, Chung CJ, Jang JH, Bae JY, Choi SR. The safety and efficacy of minimal-flow desflurane anesthesia during prolonged laparoscopic surgery. Korean J Anesthesiol. 2012 Dec;63(6):498-503. doi: 10.4097/kjae.2012.63.6.498. Epub 2012 Dec 14. PMID 23277809
- See also: Effects of Low-Flow Sevoflurane Anesthesia on Pulmonary Functions in Patients Undergoing Laparoscopic Abdominal Surgery — https://pubmed.ncbi.nlm.nih.gov/27413741/
- See also: The safety and efficacy of minimal-flow desflurane anesthesia during prolonged laparoscopic surgery — https://pubmed.ncbi.nlm.nih.gov/23277809/